CLINICAL TRIAL: NCT05882162
Title: Conventional Coronectomy vs Coronectomy in Combination Vital Pulp Treatment Using Calcium Silicate ?: A Randomized Controlled Trial up to 1 Year
Brief Title: Conventional Coronectomy vs Coronectomy in Combination Vital Pulp Treatment Using Calcium Silicate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: zeynep cukurova yilmaz (Other)
Responsible Party: Sponsor-Investigator, zeynep cukurova yilmaz, Asst. Prof. Zeynep Çukurova Yılmaz, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 66291034-604.01.01-E.46464-17
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Impacted Third Molar Tooth
Keywords: coronectomy; vital pulp therapy; impacted third mandibular molar
MeSH Terms: interventions — Dental Pulp Capping; calcium silicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): A scalpel number 15 was used to raise a triangular or envelope-shaped full-thickness mucoperiosteal flap. The bone in the buccal cavity of the third molar was removed with steel rounds and fissure burs to reach the cementum-enamel boundary. 3/4 of the tooth was cut bucco-lingually from 1-2 mm apical to the enamel cement border with the help of a high-speed surgical handpiece with a fissure steel bur. The root surface was positioned 2-3 mm apically from the surrounding alveolar bone level with the help of a steel round bur. The remaining enamel tissue and pulpal tissue in the coronal part were completely removed. Calcium silicate material was not used for pulp capping of the root pulp. During the procedure, the mandibular second molar's surface was curetted, and the surgical area was rinsed with saline solution to remove any potential surgical debris. The required number of simple sutures were used to close the surgical field without tension.
  Interventions: Procedure: Coronectomy
- Test Group (Experimental): A scalpel number 15 was used to raise a triangular or envelope-shaped full-thickness mucoperiosteal flap. The bone in the buccal cavity of the third molar was removed with steel rounds and fissure burs to reach the cementum-enamel boundary. 3/4 of the tooth was cut bucco-lingually from 1-2 mm apical to the enamel cement border with the help of a high-speed surgical handpiece with a fissure steel bur. The root surface was positioned 2-3 mm apically from the surrounding alveolar bone level with the help of a steel round bur. The remaining enamel tissue and pulpal tissue in the coronal part were completely removed. Calcium silicate material was used for pulp capping of the root pulp. During the procedure, the mandibular second molar's surface was curetted, and the surgical area was rinsed with saline solution to remove any potential surgical debris. The required number of simple sutures were used to close the surgical field without tension.
  Interventions: Procedure: Coronectomy; Procedure: Pulp Capping with calcium silicate

INTERVENTIONS:
Procedure: Coronectomy — Removal of crown part of the mandibular third molar
Procedure: Pulp Capping with calcium silicate — Application of a pulp capping material (BiodentineTM, Septodont, St Maur-des-Fosses, France) on pulp tissue to preserve the vitality of the residual pulp and prevent inflammation
  Arms: Test Group

SUMMARY:
The aim of this study was to compare the conventional coronectomy and the combined coronectomy technique with vital pulp treatment. The primary outcome of the study was to evaluate the success rates of two treatment techniques based on clinical and radiologic observations regarding inferior alveolar nerve injury, root exposure and formation of periapical lesion. The secondary outcome was to evaluate the change in periodontal condition of the second molar adjacent to the operation area, dentin bridge formation and root migration.

Between March 2018 and February 2022 eligible patients attended University Hospital for the removal of lower third molar with risk of inferior alveolar nerve (IAN) damage invited to the study. 60 teeth meeting the inclusion criteria in 52 participants were randomized to Test (with BiodentineTM, n=30) and Control (without BiodentineTM, n=30) groups. Neurological injury and post-operative pain were clinically evaluated at 12th months and 1st week, respectively. Root migration, dentin bridge formation and periapical lesion development were evaluated using Cone Beam Computed Tomography (CBCT) at 12th month. The change in the periodontal status of second molar was evaluated by measurement of pocket depth at 1st, 3rd and 12th months and the distance between base of the bone defect and the marginal crest and cemento-enamel junction and at 6th and 12th months month.

DETAILED DESCRIPTION:
The surgical removal of mandibular third molar teeth is one of the most frequently performed oral surgical procedures. One of the complications might occur during surgical removal of these teeth is injury to inferior alveolar nerve (IAN) which may lead to altered or loss of sensation to lower lip, chin, teeth and gingiva on the operated side. The risk for IAN injury may not be avoidable, even though the surgery was performed by an experienced surgeon and the positional relationship between the mandibular third molar and IAN was assessed accurately prior to surgery.

Pericoronitis, dental caries and periodontal disease are the most common pathologies associated with mandibular third molar teeth. Theoretically, removal of crown part of the teeth with a vital pulp and leaving the roots behind might be adequate to relive clinical symptoms arise from these pathologies. This technique was first described by Ecuyer and Debien in 1984 as coronectomy to prevent injury in case of close relationship of mandibular third molar with inferior IAN.

As shown previously in randomized clinical trials, fewer complications in terms of post-operative pain, IAN deficiency and dry socket were observed after coronectomy. Systematic reviews have confirmed that incidence of IAN injury was lower with coronectomy when compared to total removal in case of the lower third molar radiographically closely related with the IAN. Nerve injury was reported to occur in up to 20% of cases temporarily and 1-4% of cases permanently after total extraction, whereas 0-5.5% of cases temporarily after coronectomy.

Radiographic assessment using panaromic radiographs is the first step for coronectomy procedure. Presence of the interruption of the white line of the mandibular canal wall, darkening around the root(s), diverging of the mandibular canal, narrowing of the mandibular canal, narrowing of the root(s) and deflection of the root(s) are the indicators of increased risk for IAN injury. In recent years, cone beam computer tomography (CBCT) scanning is widely used method for further investigation to demonstrate the three-dimensional relationship between the tooth and IAN. Additionally, eligibility of the third molar for coronectomy should also be evaluated to be free of caries, pulpal inflammation and abnormal surrounding tissue. Coronectomy is contraindicated for non-compromised patients with good healing potential due to medical conditions such as diabetics, long-term steroid use, chemotherapy or radiotherapy.

One of the possible complications after coronectomy is migration and eruption of the roots left in the bone. Bone formation over the retained roots is expected to avoid eruption of these roots in the oral cavity. In case of eruption, remaining roots should be extracted. Another possible complication is periapical lesion development due to necrosis of the pulp. With conventional coronectomy procedure, no pulp treatment of the remaining roots is performed. Previous in vivo studies demonstrated that pulp retained vital after coronectomy. However, presence of pain and infection after coronectomy was reported in randomized clinical trials. Vital pulp treatment of the remaining roots with a bioactive material may have the potential to enhance both dentin and bone formation leading to reduced complications related with periapical inflammation and tooth migration.

In the literature, there is no study concerned with the clinical success of coronecyomy in combination with vital pulp treatment, except a case report. Therefore, the aim of this randomized clinical trial was to compare clinical success of conventional coronectomy and coronectomy in combination with vital pulp treatment based on clinical and radiologic evalutions. The null hypothesis tested in this study was that application of calcium silicate (Biodentine, Septodont, St Maur-des-Fosses, France) after coronectomy had no benefits to reduce above mentioned post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* - Patients without any systemic disorders
* Close relationship of the lower third molar and inferior alveolar nerve (IAN) on orthopantomography (OPTG) and Cone Beam Computed Tomography (CBCT)
* Pericoronitis around the third molar
* Caries presence or risk for caries development on the distal surface of adjacent second molar
* Follicle enlargement of less than 3 mm around the crown of the mandibular third molar on OPTG
* Teeth with complete apex development

Exclusion Criteria:

* -Presence of active infection (irreversible pulpitis) and/or pathology in the tooth
* In the presence of mobility in tooth
* Teeth with a horizontal position that are closely related to the IAN at the coronal portion
* Teeth undergoing resorption
* Smokers
* Patients who declined to take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Presence of inferior alveolar nerve injury (yes/no) | 12 months
  Hypoesthesia/hyperesthesia/dysesthesia in the lower lip or mental region of the operated side were the clinical findings for nerve injury
Root exposure (yes/no) | 12 months
  Total removal of the residual roots was required in case of eruption of the residual roots detected clinically
Periapical lesion (yes/no) | 12 Months
  Detection of periapical lesion due to necrosis of the residual root pulp radiographically (panoramic radiographs and CBCT) indicated failure of the treatment

SECONDARY OUTCOMES:
Dentin bridge formation (yes/no) | 12 months
  Presence of dentin bridge formation at the coronal part of the root pulp indicated preservation of the vitality of the root pulp
Pain (1-10) | 1 week
  Assessment of postoperative pain using a visual analog scale (VAS) printed on paper ranging from no pain to unbearable pain (1-10).
Root migration (yes/no) | 12 months
  The movement of the residual roots after coronectomy evaluated by comparing the distance between the roots with and the inferior alveolar nerve radiographically. At baseline the roots of all of the third molars were close proximity with the inferior alveolar nerve.
Maintenance of periodontal status of the adjacent tooth (yes/no) | 3,6 and 12 months
  Periodontal health of the second molar adjacent to operation site was evaluated according to measurement (milimeter) of probing pocket depth; the distance between base of the bone defect and the marginal crest and the distance between base of the bone defect and cemento-enamel junction. The measurements taken in the designated follow-ups were compared to baseline measurements to assess the change in the periodontal status.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Çukurova Yılmaz, DDS,PhD, Study Director — Private Practice
Locations (1):
- İstanbul Medipol University, Istanbul, Esenler, Turkey (Türkiye)

REFERENCES:
- [Background] Ali AS, Benton JA, Yates JM. Risk of inferior alveolar nerve injury with coronectomy vs surgical extraction of mandibular third molars-A comparison of two techniques and review of the literature. J Oral Rehabil. 2018 Mar;45(3):250-257. doi: 10.1111/joor.12589. Epub 2017 Dec 11. PMID 29171914
- [Background] Leung YY, Cheung LK. Safety of coronectomy versus excision of wisdom teeth: a randomized controlled trial. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Dec;108(6):821-7. doi: 10.1016/j.tripleo.2009.07.004. Epub 2009 Sep 26. PMID 19782621
- [Background] Renton T, Hankins M, Sproate C, McGurk M. A randomised controlled clinical trial to compare the incidence of injury to the inferior alveolar nerve as a result of coronectomy and removal of mandibular third molars. Br J Oral Maxillofac Surg. 2005 Feb;43(1):7-12. doi: 10.1016/j.bjoms.2004.09.002. PMID 15620767
- [Background] Lopes V, Mumenya R, Feinmann C, Harris M. Third molar surgery: an audit of the indications for surgery, post-operative complaints and patient satisfaction. Br J Oral Maxillofac Surg. 1995 Feb;33(1):33-5. doi: 10.1016/0266-4356(95)90083-7. PMID 7718526
- [Background] Leung YY, Cheung LK. Long-term morbidities of coronectomy on lower third molar. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Jan;121(1):5-11. doi: 10.1016/j.oooo.2015.07.012. Epub 2015 Jul 22. PMID 26337212
- [Background] O'Riordan BC. Coronectomy (intentional partial odontectomy of lower third molars). Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Sep;98(3):274-80. doi: 10.1016/S1079210404000496. PMID 15356463
- [Background] Pitros P, O'Connor N, Tryfonos A, Lopes V. A systematic review of the complications of high-risk third molar removal and coronectomy: development of a decision tree model and preliminary health economic analysis to assist in treatment planning. Br J Oral Maxillofac Surg. 2020 Nov;58(9):e16-e24. doi: 10.1016/j.bjoms.2020.07.015. Epub 2020 Aug 14. PMID 32800608
- [Background] Long H, Zhou Y, Liao L, Pyakurel U, Wang Y, Lai W. Coronectomy vs. total removal for third molar extraction: a systematic review. J Dent Res. 2012 Jul;91(7):659-65. doi: 10.1177/0022034512449346. Epub 2012 May 23. PMID 22622663
- [Background] Kohara K, Kurita K, Kuroiwa Y, Goto S, Umemura E. Usefulness of mandibular third molar coronectomy assessed through clinical evaluation over three years of follow-up. Int J Oral Maxillofac Surg. 2015 Feb;44(2):259-66. doi: 10.1016/j.ijom.2014.10.003. Epub 2014 Nov 8. PMID 25457826
- [Background] Monaco G, Vignudelli E, Diazzi M, Marchetti C, Corinaldesi G. Coronectomy of mandibular third molars: A clinical protocol to avoid inferior alveolar nerve injury. J Craniomaxillofac Surg. 2015 Oct;43(8):1694-9. doi: 10.1016/j.jcms.2015.07.006. Epub 2015 Jul 29. PMID 26321069
- [Background] Kouwenberg AJ, Stroy LP, Rijt ED, Mensink G, Gooris PJ. Coronectomy of the mandibular third molar: Respect for the inferior alveolar nerve. J Craniomaxillofac Surg. 2016 May;44(5):616-21. doi: 10.1016/j.jcms.2016.01.025. Epub 2016 Feb 18. PMID 26976696
- [Background] Tantanapornkul W, Okouchi K, Fujiwara Y, Yamashiro M, Maruoka Y, Ohbayashi N, Kurabayashi T. A comparative study of cone-beam computed tomography and conventional panoramic radiography in assessing the topographic relationship between the mandibular canal and impacted third molars. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Feb;103(2):253-9. doi: 10.1016/j.tripleo.2006.06.060. Epub 2006 Sep 1. PMID 17234544
- [Background] Gleeson CF, Patel V, Kwok J, Sproat C. Coronectomy practice. Paper 1. Technique and trouble-shooting. Br J Oral Maxillofac Surg. 2012 Dec;50(8):739-44. doi: 10.1016/j.bjoms.2012.01.001. Epub 2012 Jan 28. PMID 22285117
- [Background] Renton T. Update on coronectomy. A safer way to remove high risk mandibular third molars. Dent Update. 2013 Jun;40(5):362-4, 366-8. doi: 10.12968/denu.2013.40.5.362. PMID 23909229
- [Background] Pogrel MA, Lee JS, Muff DF. Coronectomy: a technique to protect the inferior alveolar nerve. J Oral Maxillofac Surg. 2004 Dec;62(12):1447-52. doi: 10.1016/j.joms.2004.08.003. PMID 15573343
- [Background] Goto S, Kurita K, Kuroiwa Y, Hatano Y, Kohara K, Izumi M, Ariji E. Clinical and dental computed tomographic evaluation 1 year after coronectomy. J Oral Maxillofac Surg. 2012 May;70(5):1023-9. doi: 10.1016/j.joms.2011.09.037. Epub 2011 Dec 30. PMID 22209102
- [Background] Casey DM, Lauciello FR. A review of the submerged-root concept. J Prosthet Dent. 1980 Feb;43(2):128-32. doi: 10.1016/0022-3913(80)90174-2. PMID 6766189
- [Background] da Fonseca TS, Silva GF, Guerreiro-Tanomaru JM, Delfino MM, Sasso-Cerri E, Tanomaru-Filho M, Cerri PS. Biodentine and MTA modulate immunoinflammatory response favoring bone formation in sealing of furcation perforations in rat molars. Clin Oral Investig. 2019 Mar;23(3):1237-1252. doi: 10.1007/s00784-018-2550-7. Epub 2018 Jul 7. PMID 29982967
- [Background] Nowicka A, Wilk G, Lipski M, Kolecki J, Buczkowska-Radlinska J. Tomographic Evaluation of Reparative Dentin Formation after Direct Pulp Capping with Ca(OH)2, MTA, Biodentine, and Dentin Bonding System in Human Teeth. J Endod. 2015 Aug;41(8):1234-40. doi: 10.1016/j.joen.2015.03.017. Epub 2015 May 29. PMID 26031301
- [Background] Kim YB, Joo WH, Min KS. Coronectomy of a lower third molar in combination with vital pulp therapy. Eur J Dent. 2014 Jul;8(3):416-418. doi: 10.4103/1305-7456.137660. PMID 25202226